CLINICAL TRIAL: NCT00624741
Title: Compassionate Use of Pergolide as Adjunctive Therapy to Levodopa/Carbidopa for Treating Parkinson's Disease
Brief Title: Compassionate Use Study of Pergolide in Patients With Parkinson's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRG-001
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Antiparkinsonian; Compassionate use
MeSH Terms: conditions — Parkinson Disease | interventions — Pergolide

INTERVENTIONS:
Drug: Pergolide — Pergolide tablets should be initiated with a daily dosage of 0.05 mg for the first 2 days. The dosage should then be gradually increased by 0.1 or 0.15 mg/day every third day over the next 12 days of therapy. The dosage may then be increased by 0.25 mg/day every third day until an optimal therapeutic dosage is achieved.
  Other Names: Permax

SUMMARY:
This compassionate use study is designed to monitor safety in patients who have been doing well on pergolide therapy, wish to continue treatment, and have not been able to tolerate alternative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease and treated successfully with pergolide in the recent past
* Attempt to taper off pergolide was unsuccessful and patient was unable to change to other forms of therapy for Parkinson's disease
* No evidence of cardiovalvular disease by echocardiogram conducted within 60 days prior

Exclusion Criteria:

* History or current diagnosis of cardiac valvulopathy
* Inability to undergo echocardiograms every 6 months while receiving pergolide
* Hypersensitivity to pergolide or other ergot derivatives

Sex: All
Age Groups: Child, Adult, Older Adult